CLINICAL TRIAL: NCT06305559
Title: A Placebo-controlled, Double-blind, Randomized, Phase 3 Study to Evaluate the Effect of Obicetrapib/Ezetimibe Fixed Dose Combination Daily on Coronary Plaque Characteristics in Participants With Atherosclerotic Cardiovascular Disease on Coronary CT Angiography (REMBRANDT Trial)
Brief Title: A CCTA Imaging Trial to Evaluate the Effect of Obicetrapib/Ezetimibe on Coronary Plaque
Acronym: REMBRANDT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OBEZ-302
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-11

CONDITIONS: Lipidemia; Coronary Artery Disease; Plaque, Atherosclerotic
MeSH Terms: conditions — Hyperlipidemias; Coronary Artery Disease; Plaque, Atherosclerotic | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind set-up; post randomization LDL values are not provided to sites (alert triggers are programmed for urgent follow-up)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obicetrapib/Ezetimibe (Experimental): obicetrapib 10 mg + ezetimibe 10 mg FDC daily
  Interventions: Drug: obicetrapib 10 mg + ezetimibe 10 mg FDC daily
- Placebo (Placebo Comparator): Placebo on top of baseline lipid modifying therapy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: obicetrapib 10 mg + ezetimibe 10 mg FDC daily — Active treatment
  Other Names: FDC
  Arms: Obicetrapib/Ezetimibe
Other: Placebo — Baseline lipid modifying therapy
  Arms: Placebo

SUMMARY:
This placebo-controlled, double-blind, randomized, Phase 3 study is being conducted in adult participants with high-risk atherosclerotic cardiovascular disease (ASCVD) who are not adequately controlled by their maximally tolerated lipid-modifying therapy, to assess the impact of the obicetrapib 10 mg + ezetimibe 10 mg FDC daily on coronary plaque and inflammation characteristics, evaluated using cardiovascular computed tomography angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

* Fasting serum LDL-C ≥70 mg/dL (≥1.81 mmol/L)
* Evaluable non-calcified plaque of at least 75 mm3 in the major epicardial coronary arteries
* BMI 18-40, inclusive
* Max tolerated lipid modifying therapy
* Estimated glomerular filtration rate ≥40 mL/min/1.73 m2

Exclusion Criteria:

* HbA1c ≥10.0% (≥0.100 hemoglobin fraction) or a fasting glucose ≥270 mg/dL (≥15.0 mmol/L) at Screening
* Contraindications for CCTA
* History of coronary artery bypass graft
* Active liver disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
• To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg fixed dose combination (FDC) daily on total non-calcified coronary atherosclerotic plaque volume (NCPV) at 18 months. | 18 months
  Total plaque comparison measured by CCTA

SECONDARY OUTCOMES:
Absolute change from baseline to 18 months in total NCPV in all major epicardial coronary arteries, as measured by CCTA, in participants treated with obicetrapib 10 mg + ezetimibe 10 mg FDC therapy compared with placebo. | 18 Months
  Total change in NCPV as measured by CCTA
Percent change from baseline to 18 months in LDL-C in participants treated with obicetrapib 10 mg + ezetimibe 10 mg FDC therapy compared to placebo. | 18 Months
  Change in LDL-C levels measured by central lab
Percent change from baseline to 18 months in non-calcified coronary atherosclerotic plaque volume in the most diseased coronary segment (NCPVMD), as measured by CCTA, in participants treated with FDC therapy vs placebo | 18 Months
  Percent change in plaque volume in most diseased coronary arteries measured by CCTA
Absolute change from baseline to 18 months in NCPVMD, as measured by CCTA, in participants treated with obicetrapib 10 mg + ezetimibe 10 mg FDC therapy compared with placebo. | 18 Months
  Absolute change in plaque volume in most diseased coronary arteries measured by CCTA
Change in perivascular fat attenuation index (FAI), FAI score and its age- and gender specific centile in the principal epicardial coronary arteries as measured by CCTA in participants treated with FDC therapy compared with placebo. | 18 Months
  Changes in coronary arterial fat composition measured by CCTA

CONTACTS AND LOCATIONS:
Locations (1):
- NGMR, Hialeah, Florida, United States

REFERENCES:
- [Derived] McCarthy CP, Ballantyne CM, Blankstein R, Budoff MJ, Ditmarsch M, Gibson CM, Kastelein JJP, Navar AM, Nicholls SJ, Ray KK, Shirodaria C, Williams MC, Januzzi JL Jr. Rationale and design of the REMBRANDT trial: A phase 3 study to evaluate the effect of obicetrapib/ezetimibe on coronary plaque characteristics. Am Heart J. 2025 Dec;290:325-338. doi: 10.1016/j.ahj.2025.07.012. Epub 2025 Jul 17. PMID 40683616